CLINICAL TRIAL: NCT02097810
Title: A Phase 1, Multicenter, Open-Label Study of Oral Entrectinib (RXDX-101) in Adult Patients With Locally Advanced or Metastatic Cancer Confirmed to be Positive for NTRK1, NTRK2, NTRK3, ROS1, or ALK Molecular Alterations
Brief Title: Study of Oral RXDX-101 in Adult Patients With Locally Advanced or Metastatic Cancer Targeting NTRK1, NTRK2, NTRK3, ROS1, or ALK Molecular Alterations.
Acronym: STARTRK-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RXDX-101-01; GO40784 (Other Grant/Funding Number: Hoffmann-La Roche)
Record Dates: First submitted 2014-03-21; First posted 2014-03-27 (Estimated); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Locally Advanced Solid Tumors; Metastatic Solid Tumors
MeSH Terms: interventions — entrectinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Entrectinib (RXDX-101) (Experimental): Oral entrectinib (RXDX-101)
  Interventions: Drug: Entrectinib

INTERVENTIONS:
Drug: Entrectinib
  Other Names: TrkA/TrkB/TrkC/ROS1/ALK inhibitor

SUMMARY:
Entrectinib (RXDX-101) is an orally available inhibitor of the tyrosine kinases TrkA (coded by the gene NTRK1), TrkB (coded by the gene NTRK2), TrkC (coded by the gene NTRK3), ROS1 (coded by the gene ROS1), and ALK (coded by the gene ALK). Molecular alterations to one or more of these targets are present in several different tumor types, including non-small cell lung cancer (NSCLC), colorectal cancer (CRC), prostate cancer, papillary thyroid cancer, pancreatic cancer, and neuroblastoma. Patients with locally advanced or metastatic cancer with a detectable molecular alteration in targets of interest may be eligible for enrollment.

Phase 1 will assess safety and tolerability of entrectinib via standard dose escalation scheme and determine the recommended Phase 2 dose. Safety and efficacy will be assessed in the dose expansion portion of the study.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of locally advanced or metastatic solid tumors that have a NTRK1, NTRK2, NTRK3, ROS1, or ALK molecular alteration.
* Measurable disease according to RECIST version 1.1.
* Prior cancer therapy is allowed, including crizotinib, ceritinib, and investigational drugs.
* Prior radiotherapy is allowed
* Patients with controlled asymptomatic central nervous system involvement are allowed.
* Resolution of all acute toxic effects (excluding alopecia) of any prior anti-cancer therapy to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.03 Grade less than or equal to 1.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 2.
* Adult patients age 18 years or older.
* Life expectancy of at least 3 months.

Key Exclusion Criteria:

* Current participation in another therapeutic clinical trial.
* Prior treatment with entrectinib.
* History of prolonged QTc interval (e.g., repeated demonstration of a QTc interval > 450 milliseconds).
* History of additional risk factors for torsade de pointes (e.g., family history of long QT syndrome).
* Known active infections (bacterial, fungal, viral including HIV positivity).
* Gastrointestinal disease (e.g., Crohn's disease, ulcerative colitis, or short gut syndrome) or other malabsorption syndromes that would impact on drug absorption.
* Known interstitial lung disease, interstitial fibrosis, or history of tyrosine kinase inhibitor-induced pneumonitis.
* Peripheral neuropathy ≥ Grade 2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2014-07-28 (Actual); Primary Completion 2020-06-02 (Actual); Study Completion 2020-06-02 (Actual)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity (DLT) | 28 days following first dose of entrectinib
  Determine dose-limiting toxicities of entrectinib.
Maximum Tolerated Dose (MTD) | 28 days following first dose of entrectinib
  Determine MTD of entrectinib
Recommended Phase 2 Dose (RP2D) | Approx. 6 months
  Determine RP2D of entrectinib.
Overall Response Rate (ORR) in Dose Expansion | Approx. 2 months
  Per RECIST v1.1 as assessed by Investigator.

SECONDARY OUTCOMES:
Plasma Concentrations of Entrectinib | Cycle 1 Days 1, 7, 14, 28
Disease Control | Approx. 2 years
  Per RECIST v1.1 as assessed by Investigator.
Duration of Response | Approx. 2 years
  Per RECIST v1.1 as assessed by Investigator.
Overall Survival (OS) | Approx. 2 years
Progression-Free Survival (PFS) | Approx. 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- United States (9):
  - UC Irvine Medical Center, Orange, California
  - University of California, San Francisco, Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University Of Colorado, Aurora, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Florida Cancer Specialists - Sarasota, Sarasota, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Tennessee Oncology, Nashville, Tennessee
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Doebele RC, Perez L, Trinh H, Martinec M, Martina R, Riehl T, Krebs MG, Meropol NJ, Wong WB, Crane G. Comparative effectiveness analysis between entrectinib clinical trial and crizotinib real-world data in ROS1+ NSCLC. J Comp Eff Res. 2021 Dec;10(17):1271-1282. doi: 10.2217/cer-2021-0131. Epub 2021 Aug 24. PMID 34427452
- [Derived] Dziadziuszko R, Krebs MG, De Braud F, Siena S, Drilon A, Doebele RC, Patel MR, Cho BC, Liu SV, Ahn MJ, Chiu CH, Farago AF, Lin CC, Karapetis CS, Li YC, Day BM, Chen D, Wilson TR, Barlesi F. Updated Integrated Analysis of the Efficacy and Safety of Entrectinib in Locally Advanced or Metastatic ROS1 Fusion-Positive Non-Small-Cell Lung Cancer. J Clin Oncol. 2021 Apr 10;39(11):1253-1263. doi: 10.1200/JCO.20.03025. Epub 2021 Mar 1. PMID 33646820
- [Derived] Drilon A, Siena S, Dziadziuszko R, Barlesi F, Krebs MG, Shaw AT, de Braud F, Rolfo C, Ahn MJ, Wolf J, Seto T, Cho BC, Patel MR, Chiu CH, John T, Goto K, Karapetis CS, Arkenau HT, Kim SW, Ohe Y, Li YC, Chae YK, Chung CH, Otterson GA, Murakami H, Lin CC, Tan DSW, Prenen H, Riehl T, Chow-Maneval E, Simmons B, Cui N, Johnson A, Eng S, Wilson TR, Doebele RC; trial investigators. Entrectinib in ROS1 fusion-positive non-small-cell lung cancer: integrated analysis of three phase 1-2 trials. Lancet Oncol. 2020 Feb;21(2):261-270. doi: 10.1016/S1470-2045(19)30690-4. Epub 2019 Dec 11. PMID 31838015
- [Derived] Doebele RC, Drilon A, Paz-Ares L, Siena S, Shaw AT, Farago AF, Blakely CM, Seto T, Cho BC, Tosi D, Besse B, Chawla SP, Bazhenova L, Krauss JC, Chae YK, Barve M, Garrido-Laguna I, Liu SV, Conkling P, John T, Fakih M, Sigal D, Loong HH, Buchschacher GL Jr, Garrido P, Nieva J, Steuer C, Overbeck TR, Bowles DW, Fox E, Riehl T, Chow-Maneval E, Simmons B, Cui N, Johnson A, Eng S, Wilson TR, Demetri GD; trial investigators. Entrectinib in patients with advanced or metastatic NTRK fusion-positive solid tumours: integrated analysis of three phase 1-2 trials. Lancet Oncol. 2020 Feb;21(2):271-282. doi: 10.1016/S1470-2045(19)30691-6. Epub 2019 Dec 11. PMID 31838007
- [Derived] Drilon A, Li G, Dogan S, Gounder M, Shen R, Arcila M, Wang L, Hyman DM, Hechtman J, Wei G, Cam NR, Christiansen J, Luo D, Maneval EC, Bauer T, Patel M, Liu SV, Ou SH, Farago A, Shaw A, Shoemaker RF, Lim J, Hornby Z, Multani P, Ladanyi M, Berger M, Katabi N, Ghossein R, Ho AL. What hides behind the MASC: clinical response and acquired resistance to entrectinib after ETV6-NTRK3 identification in a mammary analogue secretory carcinoma (MASC). Ann Oncol. 2016 May;27(5):920-6. doi: 10.1093/annonc/mdw042. Epub 2016 Feb 15. PMID 26884591
- [Derived] Farago AF, Le LP, Zheng Z, Muzikansky A, Drilon A, Patel M, Bauer TM, Liu SV, Ou SH, Jackman D, Costa DB, Multani PS, Li GG, Hornby Z, Chow-Maneval E, Luo D, Lim JE, Iafrate AJ, Shaw AT. Durable Clinical Response to Entrectinib in NTRK1-Rearranged Non-Small Cell Lung Cancer. J Thorac Oncol. 2015 Dec;10(12):1670-4. doi: 10.1097/01.JTO.0000473485.38553.f0. PMID 26565381